CLINICAL TRIAL: NCT07351526
Title: Inpatient Post-Acute Rehabilitation For Patients in the Midwest: a Prospective Cohort Study of Clinical Characteristics and Process Outcomes
Status: Recruiting | Type: Observational
Sponsor: University of Limerick (Other)
Responsible Party: Sponsor
Other Study IDs: 0164
Record Dates: First submitted 2025-12-08; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-10

CONDITIONS: Rehabilitation; Frailty; Complex Patients in Rehabilitation Phase
Keywords: rehabilitation; complexity; rehabilitation outcomes
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Rehabilitation improves health outcomes, reduces disability and improves quality of life. There is a significant and emerging body of international evidence to support the benefit and cost effectiveness of specialist rehabilitation services within a modern health service. The demand for rehabilitation services is growing with changes in populations and with the advances in health care and new interventions and technology.

Our overall aim is to explore the outcomes and clinical characteristics of adults who are admitted to a rehabilitation hospital in the Midwest region of Ireland during admission, at the time of their discharge and at 6 months.

DETAILED DESCRIPTION:
Rehabilitation is a dynamic and critical component of the therapeutic continuum and one that is essential if patients are to regain or maintain their life roles, health status and quality of life after serious illness or injury.

The World Health Organisation (WHO) recommends in its definition that priority is given to ensure access, for those in need, to appropriate, timely, affordable and high-quality rehabilitation interventions.

Life expectancy is improving and the population of older persons is growing with increased demand for specialist rehabilitation services. This population is at increased risk for functional decline and increased demand for healthcare services. With older adults accounting for up to 24% of all ED attendees and an anticipated rise in this number, this places increased strain on the healthcare system

The aim of this study is to establish the demographic and clinical characteristics of adults in the Midwest referred, assessed and treated in St Ita's Rehabilitation Hospital in the Mid- West of lreland.

This study will inform on resource requirements of our rehabilitation facilities to ensure that the complexity of the patients are matched by the resources provided. We will also explore the benefits of rehabilitation across a broad range of conditions and evaluate the outcomes for patients including patient reported measures.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 and over and admitted to a relevant rehabilitation unit with capacity to provide consent for inclusion.

Exclusion Criteria:

* Pregnant women and patients who are deemed not to have capacity to consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adults admitted to St Ita's Rehabilitation Hospital from February 2025 to February 2026 (inclusive) will be considered eligible for participation in the study, if they meet the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-02-22 (Actual); Primary Completion 2026-09-22 (Estimated); Study Completion 2026-09-22 (Estimated)

PRIMARY OUTCOMES:
Incidence of functional decline | Baseline
  The number of participants who experience functional decline or do not as measured by the Barthel Index (BI). Functional decline is defined as a net decrease in the number of activities of daily living performed independently as measured by the self-reported BI. The sum of all of the 10 subscales of the BI ranges from 0-20 points where a higher score indicates increased independence.
Incidence of functional decline | From the date on inception into the study until the date of discharge from hospital, assessed up to 6 months
  The number of participants who experience functional decline or do not as measured by the Barthel Index (BI). Functional decline is defined as a net decrease in the number of activities of daily living performed independently as measured by the self-reported BI. The sum of all of the 10 subscales of the BI ranges from 0-20 points where a higher score indicates increased independence.
Incidence of Functional Decline | 6 Months
  The number of participants who experience functional decline or do not as measured by the Barthel Index (BI). Functional decline is defined as a net decrease in the number of activities of daily living performed independently as measured by the self-reported BI. The sum of all of the 10 subscales of the BI ranges from 0-20 points where a higher score indicates increased independence.

SECONDARY OUTCOMES:
Healthcare use | 6 Months
  Number of services that participants were in receipt of following discharge from rehabilitation services including; GP visits, unplanned Emergency Department attendance, Outpatient appointments.
Polypharmacy level | Baseline
  Potentially inappropriate prescribing (PIP) and potentially omitted medications (POM) using the STOP START criteria. The STOPP/START Screening tools are based on the STOPP/START Prescription criteria which consist of a set of inappropriate combinations of medicines and disease (STOPP) and a set of recommended treatments for given conditions (START). There are 80 STOPP and 34 START criteria and they are grouped by physiological system e.g. cardiovascular.
Polypharmacy level | From the date on inception into the study until the date of discharge from hospital, assessed up to 6 months
  potentially inappropriate prescribing (PIP) and potentially omitted medications (POM) using the STOP START criteria. The STOPP/START Screening tools are based on the STOPP/START Prescription criteria which consist of a set of inappropriate combinations of medicines and disease (STOPP) and a set of recommended treatments for given conditions (START). There are 80 STOPP and 34 START criteria and they are grouped by physiological system e.g. cardiovascular.
Polypharmacy level | 6 Months
  potentially inappropriate prescribing (PIP) and potentially omitted medications (POM) using the STOP START criteria. The STOPP/START Screening tools are based on the STOPP/START Prescription criteria which consist of a set of inappropriate combinations of medicines and disease (STOPP) and a set of recommended treatments for given conditions (START). There are 80 STOPP and 34 START criteria and they are grouped by physiological system e.g. cardiovascular.
Frailty | From the date on inception into the study until the date of discharge from hospital, assessed up to 6 months
  Participants will be reviewed at time of discharge from rehabilitation services as to level of frailty using both the clinical frailty scale (CFS) and the identification of seniors at risk (ISAR) frailty screening tools. Both the clinical frailty scale and identification of seniors at risk were recorded at admission and again at discharge to evaluate change in frailty status over the hospital stay. The combination of tools will aim to enable examination of how initial risk screening interacts with frailty status to influence long-term functional trajectories. Higher scores on both the clinical frailty scale and identification of seniors at risk indicate higher levels of frailty and are often associated with worse outcomes. The clinical frailty scale is a 9 point rating scale (1-9) with 9 indicating the highest level of frailty (terminally ill), the identification of seniors at risk is a 6 item screening tool with a score of 2 or greater indicating increased risk of frailty.
Frailty | 6 months
  Participants will be reviewed at time of discharge from rehabilitation services as to level of frailty using both the clinical frailty scale (CFS) and the identification of seniors at risk (ISAR) frailty screening tools. Both the Clinical frailty scale and Identification of seniors at risk were recorded at 6 month follow up to evaluate change in frailty status over the hospital stay. The combination of tools will aim to enable examination of how initial risk screening interacts with frailty status to influence long-term functional trajectories. Higher scores on both the clinical frailty scale and identification of seniors at risk indicate higher levels of frailty and are often associated with worse outcomes. The clinical frailty scale is a 9 point rating scale (1-9) with 9 indicating the highest level of frailty (terminally ill), the identification of seniors at risk is a 6 item screening tool with a score of 2 or greater indicating increased risk of frailty.
Quality of life (EuroQoL-5 dimension 5 level questionnaire) | Baseline
  A questionnaire to evaluate participants health-related quality of life, assessing five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Higher scores indicate higher perception of health related quality of life. Index score (0-1) with 1 being the best and visual analogue scores (0-100) with 100 being the highest rating of overall health.
Quality of life (EuroQoL-5 dimension 5 level questionnaire) | From the date on inception into the study until the date of discharge from hospital, assessed up to 6 months
  A questionnaire to evaluate participants health-related quality of life, assessing five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Higher scores indicate higher perception of health related quality of life. Index score (0-1) with 1 being the best and visual analogue scores (0-100) with 100 being the highest rating of overall health.
Quality of life (EuroQoL-5 dimension 5 level questionnaire) | 6 Months
  A questionnaire to evaluate participants health-related quality of life, assessing five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Index score (0-1) with 1 being the best and visual analogue scores (0-100) with 100 being the highest rating of overall health.
Nursing Home Admission | 6 Months
  Number of participants who were admitted to a nursing home or residential care facility following discharge from rehabilitation services.
Mortality | 6 Months
  The number of participants who died following discharge from rehabilitation services.
Falls | 6 Months
  Number of falls sustained post discharge from rehabilitation services.

CONTACTS AND LOCATIONS:
Locations (1):
- School of Allied Health, University of Limerick, Limerick, Munster, Ireland

IPD SHARING:
Plan to Share IPD: Yes
Individual patient data collected during this study may be shared with approved researchers for the purpose of future research projects. Any data shared will be fully anonymised prior to release, with all direct and indirect identifiers removed to ensure that no participant can be identified. Only anonymised datasets will be made available, and these will be shared securely and solely for ethically approved research purposes.

REFERENCES:
- [Background] Zhang S, Lin D, Wright ME, Swallow N. Acute Inpatient Rehabilitation Improves Function Independent of Comorbidities in Medically Complex Patients. Arch Rehabil Res Clin Transl. 2022 Jan 12;4(2):100178. doi: 10.1016/j.arrct.2022.100178. eCollection 2022 Jun. PMID 35756989
- [Background] Wang H, Camicia M, DiVita M, Mix J, Niewczyk P. Early inpatient rehabilitation admission and stroke patient outcomes. Am J Phys Med Rehabil. 2015 Feb;94(2):85-96; quiz 97-100. doi: 10.1097/PHM.0000000000000226. PMID 25569470
- See also: Irish Society of physicians in Geriatric medicine strategy for rehabilitation for older people in Ireland — http://ispgm.ie/wp-content/uploads/2024/04/A-strategy-for-rehabilitation-for-older-people-in-Ireland_ISPGM_V03_web.pdf
- See also: Post-Acute Inpatient Rehabilitation Service Provision: A National Overview of HSE Funded Services — https://www.hse.ie/eng/about/who/cspd/ncps/stroke/resources/post-acute-inpatient-rehab-service-provision-a-national-overview-of-hse-funded-services-full-report.pdf
- See also: World Health Organisation fact sheet - rehabilitation — https://www.who.int/news-room/fact-sheets/detail/rehabilitation